CLINICAL TRIAL: NCT03719092
Title: Single, High Dose Vitamin A Replacement in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: High Dose Vitamin A in Preventing Gastrointestinal GVHD in Participants Undergoing Donor Stem Cell Transplant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Hannah Choe, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-18078; NCI-2018-01838 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient
MeSH Terms: interventions — Vitamin A; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Cohort (vitamin A compound) (Experimental): Participants receive vitamin A compound PO or enterally once prior to stem cell transplant.
  once over a given 24 hour period with or without food. We will re-dose at 2000 IU/kg (maximum 120,000 IU) if Week 2 Vitamin A levels remain within 10% of baseline Vitamin A.
  Interventions: Dietary Supplement: Vitamin A Compound
- Control Cohort (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Dietary Supplement: Vitamin A Compound — Given PO or enterally
  Other Names: A 313; Anti-Infective Vitamin; Antixerophthalmic Vitamin; Aquasol A; Arovit; Avibon; Avitol; Axerol; Axerophthol; Axerophtholum; Biosterol; Biovit-A; Del-Vi-A; Ido A 50; Idrurto A; Lard Factor; Lard-Factor; Ledovit A; Micelle A; Mulsal A Megadosis; Oleovitamin A; Ophthalamin; Pedi-Vit-A; Retinol, all trans-; Rinocusi Vitaminico; Vitamin A; Vitamin A Alcohol; Vitamin A USP; Vitamin A1; Vitaminoftalmina; Vitaminum A; Vogan
  Arms: Treatment Cohort (vitamin A compound)
Other: Best Practice — Receive usual care
  Other Names: Standard of care; standard therapy
  Arms: Control Cohort (usual care)

SUMMARY:
This phase I trial studies the side effects and how well high dose vitamin A works in preventing gastrointestinal graft versus host disease (GVHD) in participants undergoing donor stem cell transplant. Vitamin A deficiency is associated with increased risk of gastrointestinal GVHD. Vitamin A regulates growth and differentiation of intestinal cells and may reduce risk of gastrointestinal GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. . To determine the biologically effective and tolerable dose (BETD) level of pretransplant single, high dose vitamin A supplementation in adult allogeneic stem cell transplant recipients.

SECONDARY OBJECTIVE:

I. To evaluate the feasibility of collecting stool and profiling the gut microbiome in relation to Vitamin A.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 cohorts.

TREATMENT COHORT: Patients receive vitamin A compound orally (PO) or enterally once prior to stem cell transplant. Patients may receive vitamin A compound PO or enterally two weeks after stem cell transplant if vitamin A levels have not improved by at least 10%.

CONTROL COHORT: Patients receive usual care.

After completion of study treatment, participants are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients planned to undergo an allogeneic stem cell transplant (SCT) with an human leukocyte antigen (HLA)-matched (unrelated or related) or 1 allele mismatched (7/8) donor or haploidentical donor who received either myeloablative or nonmyeloablative conditioning for hematologic malignancies are eligible

Exclusion Criteria:

* Vitamin A hypersensitivity or allergy
* Abnormal liver enzymes outside of the institutional laboratory normal range within 30 days of screening
* Abnormal total, indirect, or direct bilirubin outside of the institutional laboratory normal range within 30 days of screening
* Enteral feeding intolerance
* Medication intolerance - history of allergic reaction to Vitamin A or other history of discontinuation to study drug due to adverse effect
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin A dose that achieves level in the upper quartile of normal range for sex in at least 2/3 cases without dose limiting toxicity | Up to day 28
  Determining a Vitamin A dose administered within 14 days prior to transplant that maintains level in the upper quartile of normal range for sex at day 28 (+/- 7 days) after stem cell infusion as well as tolerable in adult allogeneic stem cell transplant recipients.
  determining a Vitamin A dose administered within 14 days prior to transplant that maintains level in the upper quartile of normal range for sex at day 28 (+/- 7 days) after stem cell infusion as well as tolerable in adult allogeneic stem cell transplant recipients.

SECONDARY OUTCOMES:
Incidence of gastrointestinal graft versus host disease | Up to day 180 after stem cell transplant
  Cumulative incidence of GI GVHD will be calculated and graphed.
Incidence of Toxicity | Up to 28 days
  The toxicity analysis will include summarization of the toxicity and tolerability will be tabulated by dose level and summarized. Severe (grade 3+) toxicities will be summarized as well by type as well as in summary format of hematologic vs. non-hematologic severe toxicity incidence.

OTHER OUTCOMES:
Compliance of Stool collection | Pre-transplant, day 0, day 14, and day 28
  Compliance rate of take-home kit completion and inpatient stool collection
Stool microbe and vitamin A correlation | Pre-transplant, day 0, day 14, and day 28
  Correlation between stool microbes and response to vitamin A supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Choe, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu